CLINICAL TRIAL: NCT06385223
Title: A Novel Individualized Connectome-guided Approach for Precision Intermittent Theta Burst Stimulation for Depression: a Double Blind, Randomized Controlled Trial
Brief Title: A Novel Individualized Connectome-guided Approach for Precision Intermittent Theta Burst Stimulation for Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mental Health, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DSRB 2023/00680
Record Dates: First submitted 2024-04-05; First posted 2024-04-25 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-06

CONDITIONS: Depression
Keywords: neuronavigated; iTBS; Accelerated; RCT
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beam F3 targeting of accelerated iTBS (Active Comparator): Patients will receive anatomically-guided (Beam F3) accelerated iTBS.
  Participants will receive an accelerated iTBS treatment delivered with a MagVenture MagPro X100 system (MagVenture A/S, Denmark) equipped with a butterfly shaped MagVenture Cool-B65 A/P coil. The treatment course is comprised of 10 treatment sessions daily for 5 consecutive workdays for a total of 50 sessions. Each iTBS session is approximately 10 minutes (depth corrected Resting Motor Threshold of 90%, 60 cycles of 10 bursts of three pulses at 50 Hz, repeated at 5 Hz; 2s on and 8s off; 1800 pulses per session; with a 50-minute interval between sessions). All iTBS sessions will be performed by staff trained and credentialed in TMS according to Singapore College of Psychiatrists guidelines.
  Interventions: Device: Beam F3 targeted accelerated iTBS
- Individualized connectome-guided accelerated iTBS (Experimental): Patients will receive individualized connectome-guided accelerated iTBS.
  Participants will receive an accelerated iTBS treatment delivered with a MagVenture MagPro X100 system (MagVenture A/S, Denmark) equipped with a butterfly shaped MagVenture Cool-B65 A/P coil. The treatment course is comprised of 10 treatment sessions daily for 5 consecutive workdays for a total of 50 sessions. Each iTBS session is approximately 10 minutes (depth corrected Resting Motor Threshold of 90%, 60 cycles of 10 bursts of three pulses at 50 Hz, repeated at 5 Hz; 2s on and 8s off; 1800 pulses per session; with a 50-minute interval between sessions). All iTBS sessions will be performed by staff trained and credentialed in TMS according to Singapore College of Psychiatrists guidelines.
  Interventions: Device: Individualized connectome-guided accelerated iTBS

INTERVENTIONS:
Device: Beam F3 targeted accelerated iTBS — Magpro X100, Axilium Cobot, Localite camera
  Arms: Beam F3 targeting of accelerated iTBS
Device: Individualized connectome-guided accelerated iTBS — Magpro X100, Axilium Cobot, Localite camera
  Arms: Individualized connectome-guided accelerated iTBS

SUMMARY:
The Investigators propose to carry out a randomized, double-blind trial to compare the clinical efficacy of an individualized connectome-guided accelerated iTBS vs an anatomically-guided (Beam F3) accelerated iTBS. The study team will recruit both inpatients and outpatients who had been referred for TMS for the treatment of depression.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years.
2. DSM-5 diagnosis of current Major Depressive Episode.
3. Montgomery-Asberg Depression Rating Scale score of 20 or more.
4. Inadequate response to an adequate trial (4 weeks) of at least one antidepressant medication.
5. Able to give informed consent.

Exclusion Criteria:

1. DSM-5 psychotic disorder
2. Drug or alcohol abuse or dependence (preceding 3 months).
3. Rapid clinical response required, e.g., high suicide risk.
4. Significant neurological disorder, which may pose increased risks with TMS, e.g., epilepsy.
5. Metal in the cranium, skull defects, pacemaker, cochlear implant, medication pump or other electronic device.
6. Pregnancy.
7. Unsuitable for MRI.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale | Baseline, immediately post treatment, 1 month and 3 months post intervention
  Clinician rated depression rating scale, Scored 0 to 60, higher scores mean worse outcome

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology (16-Item) (Self-Report) | Baseline, daily during treatment (5 days), immediately post treatment, 1 month and 3 months post intervention
  Participant rated depression rating scale, scored 0-27, higher scores mean worse outcome
Montreal Cognitive Assessment (MoCA) | Baseline, immediately post treatment, 1 month and 3 months post intervention
  global cognitive functioning, scored 0-30, higher score means better outcome
EQ-5D (EuroQol) | Baseline, immediately post treatment, 1 month and 3 months post intervention
  Quality of life scales, scored 0-100, higher scores mean better outcome
Quality of Life Enjoyment and Satisfaction Questionnaire Short form (Q-LES-QS-SF) | Baseline, immediately post treatment, 1 month and 3 months post intervention
  Quality of life scales, scored 14-70, higher score means better outcome

OTHER OUTCOMES:
TMS induced changes in resting-fMRI functional connectivity | Baseline, immediately post treatment
  The investigators will also perform additional exploratory posthoc analyses by analysing brain imaging changes before and after TMS

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Mental Health, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No